CLINICAL TRIAL: NCT06565533
Title: A Randomized Controlled Trial Was Conducted With Participants Divided Into Three Groups: RETI, VR, and a Control Group. The RETI Group Visualized Successful FT Scenarios, the VR Group Practiced FTs in a Simulated Game Environment, and the Control Group Continued Regular Practice. Measurements Were Taken Before and After the Interventions Using Standard FT Performance Tests and the FTSE Questionnaire. Statistical Analyses, Including Mixed Factorial ANOVA, Were Performed to Evaluate the Effectiveness of the Interventions.
Brief Title: Exploring the Synergistic Effects of Virtual Reality and Retrogressive Imagery on Basketball Free Throw Performance and Self-efficacy Among University Students: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wu Jiarun (Other)
Responsible Party: Sponsor-Investigator, Wu Jiarun, Principal Investigator, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USM/JEPeM/22050298
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: RETI; VR; FTSE
Keywords: RETI; VR; FTSE; university students

STUDY DESIGN:
Intervention Model Description: The 45 students were randomly selected from South China Normal University. Of these selected students, 15 were randomly assigned to Intervention Group 1 (RETI), 15 to Intervention Group 2 (VR), and the remaining 15 to the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrogressive imagery (RETI) (Experimental): RETI protocol was implemented over eight weeks, gradually simplifying the imagery script to focus on essential aspects of the free-throw (FT) shooting technique.
  Interventions: Behavioral: Retrogressive imagery (RETI); Behavioral: Virtual Reality (VR)
- Virtual Reality (VR) (Experimental): Using Virtual Reality (VR) technology, participants are fully immersed in an intense basketball game experience.
  Interventions: Behavioral: Retrogressive imagery (RETI); Behavioral: Virtual Reality (VR)

INTERVENTIONS:
Behavioral: Retrogressive imagery (RETI) — Week 1-2: Participants were asked to imagine a complete version of the FT imagery script included: a) Visualizing the court lines, the basket, and themselves standing at the free-throw line, focusing on their shooting technique. b) Imagining teammates and opponents positioned around the key, noting the main colors in the scene c) Imagining the coach standing on the sideline encouraging them, and paying attention to the sounds of the audience and the cheers from a close friend in the stands. d) Visualizing a high-pressure situation, experiencing the emotions felt during a real game with one second left on the clock, trailing by one point, with the game's outcome depending on their FT shot. Week 3-4: The exception of content "d"from the full script. Week 5-6: The exception of content "c""d"from the full script. Week 7-8: The exception of content "b""c""d"from the full script.
Behavioral: Virtual Reality (VR) — Standing on a lifelike full-sized basketball court, they observe smooth flooring and clear markings. Teammates and opponents don variously colored uniforms, while referees stand ready at the sidelines. Referees position teammates and opponents around the basket as participants feel the texture and weight of the basketball in their hands, as if gripping it for real. The sounds of cheering spectators and encouraging shouts from teammates and coaches further enhance their focus. Participants adjust their stance, noticing beads of sweat trickling down their arms as they prepare for the FT. With bent knees, they ready themselves for the shot, exerting every ounce of their strength as the ball leaves their hands and soars towards the basket. As the ball accurately swishes through the net, the crowd erupts into thunderous applause, and the scoreboard's change in score brings an overwhelming sense of joyous victory.

SUMMARY:
This research contributes to the growing body of evidence supporting the use of mental training techniques in sports. By demonstrating the effectiveness of RETI and VR in improving FT performance and FTSE, this study provides valuable insights for coaches, athletes, and sports psychologists.

ELIGIBILITY:
Inclusion Criteria:

participants to be university students aged 17 to 23 years, with the ability to read and communicate in Mandarin.

Exclusion Criteria:

students with visual, auditory, or other motor impairments

Ages: 17 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Free Throw (FT) Shooting Performance | week 8
  Free throw (FT) are a closed skill technique used for scoring points under practice, field study, or game conditions. Testing was conducted before, during, and after the intervention. FTs are typically awarded to players who are fouled while shooting, and the player takes the shot from behind the FT line, which is 15 feet away from the basket. Each successful FT is worth one point. In this study, to measure shooting accuracy more precisely, we employed the following scoring system: a shot that goes through the basket without touching the rim scores 3 points; a shot that goes in after hitting the rim scores 2 points; a shot that hits the rim but does not go in scores 1 point; and a complete miss scores 0 points. Each testing session comprised two sets of 10 FT shots, with a 15-minute rest period between the sets. The total score for each testing session was calculated by summing the scores from the two sets of 10 shots, resulting in a possible range of 0 to 60.
Free throw shooting self-efficacy (FTSE) | week 8
  We utilized the Free-Throw Self-Efficacy (FTSE) scale developed by Fazel (2015) to measure participants' self-efficacy in basketball free-throw shooting, following the microanalytic technique guidelines proposed by Bandura (2006). Participants were asked to imagine taking 10 consecutive free throw and to rate their confidence in successfully making each of these shots. Specifically, they were asked to indicate how certain they were that they could successfully make 1 out of 10, 2 out of 10, and so on, up to 10 out of 10 free throw. Participants rated their confidence on a scale from 0 (completely uncertain) to 10 (very certain).

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia